CLINICAL TRIAL: NCT03772691
Title: Lateral Suspension Versus Sacropexy for Treatment of Apical Pelvic Organ Prolapse
Brief Title: Lateral Suspension and Sacropexy for Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal M.fekry, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSS
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lateral suspension (Experimental): All operations will be performed with patient in loyd davies position, sterilization of the perineum then sterilization of the vagina
  Interventions: Procedure: lateral suspension
- sacropexy (Active Comparator): Our ﬁrst passage is the peritoneum incision overlying the sacral promontory (L5-S1) to expose the anterior longitudinal ligament, which is the anchorage point of the mesh on the sacrum. We create a tunnel under the peritoneum on the right side through the cul-de-sac of Douglas till reach the cervix or vaginal cuff (after hysterectomy).
  Interventions: Procedure: sacropexy

INTERVENTIONS:
Procedure: lateral suspension — • The vesico-vaginal space was found between the bladder and the anterior vaginal wall in the fascia plane. A polypropylene mesh (25 , 25 cm, Ethicon, Inc., Somerville, NJ) was cut to obtain two long arms (15-20 mm wide) and a rectangular piece (4-7 cm wide).
  Arms: lateral suspension
Procedure: sacropexy — • The mesh is fixed on the anterior longitudinal ligament of sacrum with separated number 1 prolene sutures. The other end of the mesh is passed through the peritoneal tunnel and fixed to the cervix using prolene 1 and vicryl o sutures.
  Arms: sacropexy

SUMMARY:
Pelvic organ prolapse (POP) is considered one of the commonest gynecologic health problems all over the world. Pelvic organ prolapse (POP) is common and can be seen in up to 50% or more of parous women. The annual aggregated rate of associated surgery for pelvic organ prolapse is in the range of 10-30 per 10,000 women. It is estimated that women have an 11-19% life-time risk of undergoing surgery for POP. This rate is projected to increase over the next 2-3 decades. Apical POP refers any descent of the cervix or the vaginal cuff scar(as after hysterectomy) below a point which is 2 cm less than the total vaginal length about the plane of the hymen. Apical POP is due to defect in apical support with damage to the cardinal and uterosacral ligaments. Apical pelvic organ prolapse is a common issue in our country with significant incidence rate due to many predisposing factors including increasing age, higher gravidity and parity (especially the number of vaginal births)

DETAILED DESCRIPTION:
By one estimate, the demand for health care services related to pelvic floor disorders will increase at twice the rate of the population itself . So we need adequate understanding of the best surgical method for treating apical POP which is accepted worldwide and also must be cost effective with least perioperative complications. Abdominal sacropexy is considered now the gold standard operation for treatment of apical pelvic organ prolapse. In this technique, the mesh is ﬁxed to the anterior longitudinal ligament at the sacral promontory. It is used either with uterine preservation (sacrohysteropexy) or after hysterectomy (sacrocolpopexy) for treatment of vault prolapse .However , many intraoperative complication can occur including hemorrhage or transfusion or both occurred in 4.4% , intestinal injury or rectal injury in 1.6% (0.4% to 2.5%),and ureteral injury in 1.0% of cases. Postoperative complications include paralytic ileus in 3.6%.transient femoral nerve injury and vertebral osteomyelitis . Also, despite that sacropexy provide good apical support, but the high prevalence of cystocele and urinary tract symptoms in patients reaches up to 8% . Consequently, it is not surprising that the majority of failures following sacrocolpopexy occur in the anterior compartment. Lateral suspension with mesh was ﬁrst reported by Dubuisson in 1998 for the treatment of pelvic organ prolapse . The lateral suspension avoids both the risk of vascular injury and nerve damage of sacrocolpopexy with success rate up to 88% of cases.

ELIGIBILITY:
Inclusion Criteria:

* Apical prolapse Stage 2-4 according to POP-Q system
* Uterine preservation or after hysterectomy
* Sexually active or not.

Exclusion Criteria:

* Pregnancy or up to 6 months postpartum.
* Current Urinary tract infection proved by urine analysis or urine culture.
* Patient unfit for surgery.
* Previous suspension operations.
* Uncontrolled diabetic patients.
* Urge incontinence.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
rate of occurance of denovo stress urinary incontinence | 18 months
  number of patients developed new onset postoperative stress urinary incontinence
The rate of Improvement of urinary symptoms | 18 months
  Improvement of symptoms using Abramsc Development and psychometric evaluation of the International consultation on incontinence and Vaginal Symptoms Questionnaire maximum score:178, minimum score:0 high score means better outcome , low score means worse outcome

SECONDARY OUTCOMES:
objective assessment of prolapse stage | 18 months
  improvement of POP-Q system postoperatively
assessment of sexual function | 18 months
  improvement of female sexual function index postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Derived] Sayed E, Mitwally A, Abdelmagied A, Fetih A, Fekry M. Transperineal Ultrasound Evaluation of Bladder Parameters in Patients with Apical Prolapse Undergoing Lateral Suspension or Sacropexy. J Obstet Gynaecol India. 2024 Apr;74(2):170-175. doi: 10.1007/s13224-023-01912-2. Epub 2023 Dec 19. PMID 38707876